CLINICAL TRIAL: NCT05640960
Title: Undifferentiated Embryonal Sarcoma of the Liver
Brief Title: Undifferentiated Embryonal Sarcoma of the Liver: Evaluation of the Relapse Profile According to the Therapies Administered
Acronym: SARCOM
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7979
Record Dates: First submitted 2022-11-28; First posted 2022-12-07 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Hepatic Sarcoma
Keywords: Embryonal Sarcoma; Embryonic Sarcoma; Hepatoblastoma; Hepatocarcinoma; Hepatic Sarcoma; Undifferentiated (Embryonal) Sarcoma
MeSH Terms: conditions — Hepatoblastoma; Carcinoma, Hepatocellular; Disorders of Sex Development; Sarcoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Undifferentiated embryonal sarcoma of the liver is the 3rd most common malignant liver tumor after hepatoblastoma and hepatocellular carcinoma with a peak incidence between 6 and 10 years of age. Historically, it is a tumor treated only by surgery with a poor prognosis. In the last decade, the combination of more intensive chemotherapy and, more randomly, radiotherapy, has significantly improved the survival rate of these patients. Due to its low incidence, there are few series reported in the literature and to date there is no specific treatment protocol for the management of these tumors.

It seems appropriate to review the management of these tumors in France in order to discuss the best therapeutic strategy.

ELIGIBILITY:
Inclusion criteria:

* Any patient aged 0 to 25 on the date of inclusion in the study
* Treatment carried out in France (included in NRSTS 2005, in the childhood cancer registry or in an SFCE center)
* Start of treatment from 01/01/2008 to 31/12/2018
* Diagnosis of undifferentiated embryonal sarcoma of the liver defined by a compatible histological analysis
* Adult subject who has not expressed, after being informed, his opposition to the reuse of his data for the purposes of this research
* Minor subject (and/or his parental authority) who has not expressed, after being informed, his opposition to the reuse of his data for the purposes of this research

Exclusion criteria:

* Refusal to participate in this research
* Diagnosis of rhabdoid tumor, rhabdomysarcomas, angiosarcomas, PNET
* Absence of histological and/or molecular documentation.

Ages: 1 Year to 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patient aged 0 to 25 with treatment carried out in France from 01/01/2008 to 31/12/2018
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Describe the relapse profile of children with undifferentiated hepatic sarcoma according to the therapies received | 3 years after treatment
  the primary endpoint is event-free survival (progression, death, relapse) at 3 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Service Pédiatrie Onco-hématologie - Pédiatrie III - CHU de Strasbourg - France, Strasbourg, France